CLINICAL TRIAL: NCT02122237
Title: Cathodal Transcranial Direct Current Stimulation in Chronic Migraine: Neurophysiological Study and Pilot Therapeutic Trial
Brief Title: Cathodal tDCS in Chronic Migraine: Neurophysiological Study and Pilot Therapeutic Trial
Acronym: CATCHROMIG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean Schoenen, Honorary Full Professor, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-1289
Record Dates: First submitted 2013-11-04; First posted 2014-04-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cathodal Cefaly tDCS (Experimental): Cathodal Cefaly tDCS is delivered over the visual cortex at 2 mA of intensity, for 20 minutes, everyday for 2 months, in 14 patients. The anode is placed over the left DLPFC.
  Interventions: Device: Cefaly tDCS

INTERVENTIONS:
Device: Cefaly tDCS — Cefaly tDCS (transcranial direct current stimulation) is able to modify cortical excitability, in particular cathodal tDCS decreases it. The side effects of tDCS are minor, especially sensations of itching and scalp paresthesias.

SUMMARY:
Cathodal tDCS decreases the excitability of the cerebral cortex and its daily application during intercritical phase, may have a therapeutic effect in chronic migraine.

DETAILED DESCRIPTION:
During the interictal phase, the cerebral cortex is characterised by a hyperresponsiveness to repeated sensory stimuli, manifested by a lack of habituation or adaptation of cortical responses. Lack of habituation has been shown in the visual cortex in studies of visual evoked potentials (VEP) during the interictal period and it is possibly explained by a reduction in the cortical pre-activation level due to thalamo-cortical dysrhythmia. Just before and during the migraine attack, cortical reactivity changes drastically: habituation is restored and the amplitude increases. In chronic migraine (headache occurring on 15 or more days per month for more than 3 months with features of migraine headache on at least 8 days per month), VEPs habituate normally like those recorded during attacks of episodic migraine, but have in addition an increased amplitude in the 1st block of responses. Chronic migraine was therefore compared to a "never ending migraine attack" accompanied by cortical hypersensitivity.

In this study the investigators aim to demonstrate that cathodal tDCS over the visual cortex with simultaneous anodal tDCS over the left dorsolateral prefrontal cortex is able: 1) to reduce cortical hypersensitivity and habituation as assessed by VEPs and contact heat evoked nociceptive potentials (CHEPS), as well as to decrease pain perception assessed by quantitative sensory testing (QST) and the nociceptive blink reflex (nBR); 2) to decrease headache and migraine frequency.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic migraine (ICHD III beta 1.3) with or without medication overuse

Exclusion Criteria:

* others diseases or contraindications to tDCS (epilepsy, pacemaker, metal prosthetics)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Migraine frequency | 6 months
  The investigators evaluate migraine frequency at baseline, during the treatment and 2 months after its end.

SECONDARY OUTCOMES:
Migraine intensity | 6 months
  The investigators evaluate migraine intensity at baseline, during the treatment and 2 months after its end.
Acute medication intake | 6 months
  The investigators evaluate acute medication intake at baseline, during the treatment and 2 months after its end.
Attack duration | 6 months
  The investigators evaluate attack duration at baseline, during the treatment and 2 months after its end.
Scores at psychological scales | 6 months
  The investigators evaluate scores at psychological scales at baseline, during the treatment and 2 months after its end.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Magis, MD,PhD, Principal Investigator — University of Liege; Jean Schoenen, MD,PhD, Study Director — University of Liege
Locations (1):
- Roberta Baschi, Liège, Belgium, Belgium